CLINICAL TRIAL: NCT06761157
Title: Transrectal Evaluation After Discoid Resection For Endometriosis Intestinal
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RESDISCO2021
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Deep Endometriosis
Keywords: endometriosis; discoid resection; deep endometriosis; intestinal
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluating the success of rectosigmoidoscopy performed after intestinal resection in women with deep endometriosis during surgery

DETAILED DESCRIPTION:
Endometriosis is an inflammatory, benign, oestrogen-dependent condition that affects 10-15% of women of reproductive age. It is characterised by the presence of endometrial tissue, glands and stroma, outside the uterine cavity. Endometriosis may present in the pelvis as superficial peritoneal, ovarian or deep infiltrating. The reported prevalence of bowel or recto-vaginal space involvement among women with endometriosis ranges from 5% to 25% (2). Surgery is the treatment of choice for deep endometriosis with bowel involvement when drug therapy alone is ineffective in treating symptoms. Surgical techniques for intestinal endometriosis can be divided into full-thickness techniques (discoid or segmental resection) and non-full-thickness techniques (shaving).

Focusing on women who underwent a discoid resection, 3.7% of 80 reported a recto-vaginal fistula and the same percentage showed early rectorrhagia requiring endoscopic treatment after surgery. In general surgery rectosigmoidoscopy has shown encouraging results as a feasible, safe and effective technique in reducing the risk of complications related to intestinal anastomosis. There are no studies in the literature evaluating the role of rectosigmoidoscopy as a routine practice in gynaecological surgery for endometriosis, so we rely on the experience of general surgeons. In particular, the lack of data does not allow us to evaluate the feasibility of rectosigmoidoscopy during deep endometriosis surgery in terms of the success of the procedure itself and the additional operative time taken. The latter aspect is also important from the point of view of health policy due to the increased cost of the operating theatre directly related to the time taken for the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 50 years
* Women with diagnosis made by instrumental examination such as transvaginal ultrasound, of deep endometriosis with suspected bowel involvement
* Women undergoing segmental or discoid resection for bowel endometriosis
* Obtaining informed consent

Exclusion Criteria:

* Patients who are candidates for elective laparotomic surgery
* Patients with concomitant inflammatory bowel disease known in history (inflammatory bowel syndrome)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with deep endometriosis with suspected bowel involvement who will undergo segmental or discoid resection for the period of one year following the date of study approval
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Success rate of rectosigmoidoscopic procedure in patients with deep endometriosis with bowel involvement undergoing segmental or discoid resection surgery | 3 months after surgery
  Ratio of the number of successfully completed interventions to the total number of interventions performed using rectosigmoidoscopy. The success of the intervention is determined following qualitative evaluation of the anastomosis

SECONDARY OUTCOMES:
Incidence of intraoperative complications: rectorrhagia, leakage, mucosal crash, intussusception, anastomosis stenosis, intraperitoneal hemorrhage, conversion to laparotomy surgery | During surgery
  Ratio of the number of procedures in which any of the intraoperative complications described above occurred to the total number of procedures using rectosigmoidoscopy
Incidence of postoperative complications within the first three months post-segmental or discoid resection surgery among patients undergoing rectosigmoidoscopy and patients undergoing the same surgery without rectosigmoidoscopy | 3 months after surgery
  Ratio of the number of surgeries in which any of the above postoperative complications occurred to the total number of surgeries using rectosigmoidoscopy
Operating time duration in patients undergoing discoid or segmental resection with or without the use of intraoperative rectosigmoidoscopy | 3 months after surgery
  Percentage difference between average surgical durations in patients undergoing resection surgery with and without a rectosigmoidoscopy procedure. Lacking baseline data, an increase, compared with patients who did not undergo rectosigmoidoscopy, of up to 20% in average surgical time is considered reasonable

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Casadio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy